CLINICAL TRIAL: NCT01774617
Title: Comparative Analysis of Indocyanine Green Clearance Test, MELD Score, MELD-Na Score, Transient Elastography and Hepatic Venous Pressure Gradient to Evaluate Prognosis of Patients on Liver Transplant Waiting List
Brief Title: Comparative Analysis of Different Tests to Evaluate Prognosis of Patients on Liver Transplant Waiting List
Status: Completed | Type: Observational
Sponsor: Guilherme Rezende (Other)
Collaborators: Rio de Janeiro State Research Supporting Foundation (FAPERJ) (Other Government)
Responsible Party: Sponsor-Investigator, Guilherme Rezende, Associate Professor, MD PhD, Universidade Federal do Rio de Janeiro
Organization: Universidade Federal do Rio de Janeiro (Other)
Other Study IDs: HHL/UFRJ-04; CAAE 06343212.8.0000.5257 (Registry Identifier: Plataforma Brasil CEP/CONEP)
Record Dates: First submitted 2013-01-22; First posted 2013-01-24 (Estimated); Last update posted 2020-10-09 (Actual); Status verified 2020-10

CONDITIONS: Cirrhosis; Liver Failure; Portal Hypertension
Keywords: portal hypertension; elastography; Hepatic venous pressure gradient measurement
MeSH Terms: conditions — Fibrosis; Liver Failure; Hypertension, Portal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients with advanced liver disease: Inclusion criteria are diagnosis of cirrhosis with portal hypertension detected by abdominal ultrasound with color Doppler flowmetry or upper digestive endoscopy. Exclusion criteria were age 18 or older, previous contrast allergy, hepatocellular carcinoma or any malignancy except basocellular carcinoma, renal failure (creatinine level >1.5 mg/dL), severe bleeding disorder (prothrombin activity test < 30% or platelets count <35,000/mcL) or decompensated cirrhosis characterized by severe ascites or grade II or higher encephalopathy. Patients with alcoholic cirrhosis should be abstinent for at least six months.

SUMMARY:
It is a cohort to evaluate the power of different diagnostic tests in predicting the prognosis of patients with severe liver disease.

Patients with decompensated liver cirrhosis on the waiting list for liver transplantation will be evaluated with comparison of different diagnostic tests according to the MELD score (Model for End-Stage Liver Disease), MELD-Na (Model for End-Stage Liver Disease and sodium), indocyanine green clearance test, hepatic venous pressure gradient and transient elastography. All patients will be submitted to all the tests and prospectively followed for 6 months, to establish mortality and complications related to liver disease in order to define the value of each method to predict outcomes.

ELIGIBILITY:
Inclusion Criteria:

* the study includes patients (80 patients)
* were male and female
* aged between 18 and 69 years with chronic liver disease
* with MELD inclusion greater than or equal to 14 to 30

Exclusion Criteria:

* they have been transplanted
* have a diagnosis of primary malignant liver (HCC) signed by imaging tests performed
* MELD scores greater than 30.

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cirrhotic patients on the liver transplantation waiting list of a single center.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2015-12 (Actual); Primary Completion 2018-11 (Actual); Study Completion 2018-11 (Actual)

PRIMARY OUTCOMES:
All cause mortality | 6 months
  Mortality within 6 months after evaluation, classifying as related or non-related to liver disease

SECONDARY OUTCOMES:
Chronic liver failure and portal hypertension complications | 6 months
  Complications:
  * gastroesophageal variceal bleeding
  * worsening of hepatic encephalopathy
  * decompensated ascites and spontaneous bacterial peritonitis
  * hepatorenal syndrome

CONTACTS AND LOCATIONS:
Overall Officials: Guilherme FM Rezende, MD PhD, Study Chair — Universidade Federal do Rio de Janeiro
Locations (1):
- Hospital Universitário Clementino Fraga Filho / Federal University of Rio de Janeiro, Rio de Janeiro, Rio de Janeiro, Brazil